CLINICAL TRIAL: NCT03725748
Title: Normal Saline Versus Betadine Use to Reduce the Incidence of Wound Infection in Cesarean
Brief Title: Normal Saline Versus Betadine Use to Reduce the Incidence of Wound Infection in Cesarean Section
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, hadeer meshal, assistant prfessor, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: assistant professor2
Record Dates: First submitted 2018-10-20; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Incidence of cs Scar Infection
Keywords: saline, betadine, cesarean scar infection
MeSH Terms: interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no irrigation group (No Intervention): nothing used for irrigation of cs scar
- saline irrigation group (Placebo Comparator): saline used for irrigation the cs scar before closure
  Interventions: Other: irrigation
- betadine irrigation group (Experimental): betadine used for irrigation of cs scar
  Interventions: Other: irrigation

INTERVENTIONS:
Other: irrigation — irrigation the edges of the cs scar before closure
  Arms: betadine irrigation group; saline irrigation group

SUMMARY:
This is a prospective randomized controlled study to the difference between using normal saline or betadine irrigation of wound prior to skin closure in reducing the incidence of wound infection after Cesarean section.

DETAILED DESCRIPTION:
This study will be conducted at the Department of Obstetrics & Gynecology, Kasr El-Ainy Teaching Hospital, Faculty of Medicine, Cairo University, from February to July 2018.

We include in our study 3oo pregnant women who will undergo Cesarean section. All participants will be divided into 3 groups with a 1:1:1 ratio with 100 patients in each group. Each participant will provide an informed written consent.

Consenting patients will be pre-operatively randomised using numerically ordered cards in sealed envelopes to either the group 1 (wound irrigation with 100 ml of normal saline before skin closure) or the group 2 (wound irrigation with 50 ml of 10% aqueous povidone iodine solution ̋ Betadinȅ ) or the control group (no wound irrigation with normal saline nor betadine).Subjects candidate for the study will be 37 weeks' gestation and require a cesarean section (elective or emergency). Patients with allergy to iodine, history of immunosuppressive drug use, gestationaldiabetes mellitus or preeclampsia, anemic patients, ruptured of membranes and feverish patients will be excluded from the study.

The primary outcome will be the incidence of wound infection. Wound infection is diagnosed when the wound drained purulent material or serosanguineous fluid in association with induration, warmth and tenderness. Suspected wound infections are opened for confirmation and wound cultures will be taken. Haematoma, seroma, or wound breakdown in the absence of the previouslydiscussed signs is not considered a wound infection.Wounds are examined twice daily during hospitalization for evidence of infection. After discharge, the women are instructed on the signs and symptoms of wound infection, and asked to contact one of the co-authors immediately if any of the listed symptoms appeared. All participants are examined at 2 and 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects candidate for the study will be 37 weeks' gestation
* require a cesarean section (elective or emergency).

Exclusion Criteria:

* Patients with allergy to iodine
* history of immunosuppressive drug use,
* gestationaldiabetes mellitus
* preeclampsia
* anemic patients
* ruptured of membranes
* feverish patients

Ages: 19 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
incidence of cs scar infection | 2 to 6 weeks
  incidence of cs scar infection

SECONDARY OUTCOMES:
incidence of hematoma, seroma | 2 to 6 weeks
  incidence of hematoma, seroma, wound breakdown

CONTACTS AND LOCATIONS:
Overall Officials: fady salah, lecturer, Study Director — Director
Locations (1):
- Kasr El Ainy, Cairo, Egypt